CLINICAL TRIAL: NCT03270371
Title: Medium-term Modulation of the Inflammatory Profile by Medium-cut Off Membranes in Patients With End Stage Renal Disease
Brief Title: Modulation of Inflammation by Medium Cut Off Membranes
Acronym: MCO-IF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MCO-CS-559/16S
Record Dates: First submitted 2017-08-25; First posted 2017-09-01 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Cardiovascular Diseases; End Stage Renal Disease
MeSH Terms: conditions — Cardiovascular Diseases; Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: Medium cut off Dialyzer compared with standard of care High-Flux Dialyzer (Fx Cor Diax 60®). No others changes in our standard of care maintenance dialysis is planned, dialysis specific parameters such as blood flow will be kept unchanged during the study period).
Masking Description: no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MCO Dialysis (Experimental): Theranova Dialyzer
  Interventions: Device: Medium cut off dialysis
- Standard High Flux Dialysis (Active Comparator): Standard High Flux Dialyzer
  Interventions: Device: Standard High Flux Dialyzer

INTERVENTIONS:
Device: Medium cut off dialysis — Hemodialysis
  Other Names: Theranova Dialyzer
  Arms: MCO Dialysis
Device: Standard High Flux Dialyzer — Hemodialysis
  Arms: Standard High Flux Dialysis

SUMMARY:
This study examines whether medium-cut off dialysis results in improved blood purification of large middle molecules e.g. inflammatory molecules compared to hemodialysis (HD) treatments with conventional high-flux dialyzers.

DETAILED DESCRIPTION:
Cardiovascular events and sepsis remain the leading causes of mortality in patients on maintenance hemodialysis. Thus expectancy of life for these patients is comparable to the prognosis of metastasized cancer. So far the exact mechanisms causing excess mortality in hemodialysis patients remain elusive, but chronic inflammation seems to play a central role in the pathogenesis of cardiovascular disease in HD patients.

Keeping this in mind the Theranova medium-cut off membrane, with its ability to clear middle molecules (0,5-50 kDa), seems suitable to further improve clearance of inflammatory mediators as the non-protein bound inflammatory mediators lie within the cut off range of this membrane. The investigators designed this study to get information on the changes in the inflammatory milieu in dialysis patients when using medium-cut off membranes which are know to significantly reduce cytokines compared to standard high-flux dialyzers.

ELIGIBILITY:
Inclusion Criteria:

* time since initiation of dialysis > 3 months
* age > 18 years

Exclusion Criteria:

* time since initiation of dialysis < 3 months
* age < 18 years
* ongoing acute or chronic infection/malignoma, because this will interfere with inflammatory baseline values
* major surgery less than 2 weeks before inclusion in the study
* pregnancy
* mental illness
* lack of written and informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2018-10 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Change in inflammation | 240 days (cross-over design, multiple measurements)
  change of inflammatory score (inflammatory score is derived from multiple biomarkers)

SECONDARY OUTCOMES:
Change in calcification status | 240 days (cross-over design, multiple measurements)
  calcification score derived from several pro- and anticalcifying biomarkers
change in calcification propensity | 240 days (cross-over design, multiple measurements)
  this values measures the resistence of serum to a calcification stimulus

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Schmaderer, MD, Principal Investigator — attending Department of Nephrology, Klinikum rechts der Isar
Locations (1):
- Department of nephrology, Klinikum rechts der Isar, München, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ronco C, La Manna G. Expanded Hemodialysis: A New Therapy for a New Class of Membranes. Contrib Nephrol. 2017;190:124-133. doi: 10.1159/000468959. Epub 2017 May 23. PMID 28535525
- [Background] Zickler D, Schindler R, Willy K, Martus P, Pawlak M, Storr M, Hulko M, Boehler T, Glomb MA, Liehr K, Henning C, Templin M, Trojanowicz B, Ulrich C, Werner K, Fiedler R, Girndt M. Medium Cut-Off (MCO) Membranes Reduce Inflammation in Chronic Dialysis Patients-A Randomized Controlled Clinical Trial. PLoS One. 2017 Jan 13;12(1):e0169024. doi: 10.1371/journal.pone.0169024. eCollection 2017. PMID 28085888